CLINICAL TRIAL: NCT03580239
Title: Placebo-Controlled, Randomized, Prospective and Multicenter Trial of Everolimus in Castrated Resistant Prostate Cancer Patients With PI3K-AKT-mTOR Signaling Pathway Deficiency
Brief Title: Everolimus in Castrated Resistant Prostate Cancer(CRPC)Patients With PI3K-AKT-mTOR Signaling Pathway Deficiency
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Tianjin First Central Hospital (Other); The Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine，China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRPC-EVE
Record Dates: First submitted 2018-06-25; First posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: CRPC; Everolimus; mTOR
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Everolimus & Best Supportive Care (Experimental): Everolimus will be administered at a dose of 10mg/day orally once a day. One cycle of therapy consists of 28 days.The patients also receive the best supportive care.
  Interventions: Drug: Everolimus
- Placebo & Best Supportive Care (Placebo Comparator): Placebo will be administered at a dose of 10mg/day orally once a day. One cycle of therapy consists of 28 days.The patients also receive the best supportive care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Everolimus — Everolimus will be treated at a dose of 10mg/day orally once a day. One cycle of therapy consists of 28 days. The patients also receive the best supportive care.
  Other Names: Novartis Pharma Schweiz AG
  Arms: Everolimus & Best Supportive Care
Drug: Placebo — Placebo will be treated at a dose of 10mg/day orally once a day. One cycle of therapy consists of 28 days. The patients also receive the best supportive care.
  Arms: Placebo & Best Supportive Care

SUMMARY:
Investigators seek a new therapeutic strategy for castrated resistant prostate cancer(CRPC) patients with PI3K-AKT-mTOR signaling pathway deficiency by next generation sequencing(NGS).

DETAILED DESCRIPTION:
The prognosis of castrated resistant prostate cancer(CRPC) is very poor.Now,there is not an ideal therapeutic strategy.Further clarifying its mechanism and finding more effective therapeutic targets on this basis are the clinical problems to be solved urgently. More and more studies have confirmed that the role of PI3K-AKT-mTOR signaling pathway in the development of castration resistance to prostate cancer.By next generation sequencing of 115 patients with CRPC, investigators found that 22% of the patients had mutations in the PI3K-AKT-mTOR signaling related genes.Investigators found that 50% of the patients could benefit from the mTOR inhibitors.But the specific clinical significance and molecular mechanism are urgently needed to be elucidated. This project is based on the hypothesis that Everolimus can target CRPC patients with PI3K-AKT-mTOR signaling pathways deficiency.So,investigators intend to peform a prospective, randomized, controlled,multicenter clinical study to find potential therapeutic targets and treatment strategies for CRPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with advanced refractory castration resistant prostate cancer(CRPC).
2. Patients with histologically or cytologically confirmed prostate cancer.
3. Conventional treatment failed advanced CRPC patients,routine treatment including:radical prostatic cancer surgery,castration, ADT, amieton /inololamine new endocrine therapy,docetaxel intravenous drug resistance, or intolerance of toxic and side effects.
4. Patients must be able to provide blood samples or tissue samples for testing. The amount of blood samples should be able to meet the requirements of DNA extraction and quality control:

   I.Sample type: DNA samples without RNA degradation and pollution free.

   II.A single sample size of more than 500 ng (using Roche library platform,Illumina sequencing platform).

   III.The sample concentration is more than 40 ng/L (using Roche building database platform; Illumina sequencing platform); IV.The purity of the sample is OD 260/280=1.8~2;
5. After next generations of sequencing, all the patients were found to have defects in the PI3K-AKT-mTOR signaling pathway, including the following molecular markers: PI3K, AKT, mTOR, PTEN, TSC1, TSC2 and so on.
6. The expected survival time is more than 4 weeks.
7. Patients with Karnofsky(KPS) functional status score > 60 and Eastern Cooperative Oncology Group(ECOG)state score 0-2 points.
8. Patients organ function level must comply with the following requirements:

   I.Hematological parameters: the absolute count of neutrophils is more than 1.5*109/L, platelets count is more than 80*109/L, hemoglobin is more than 9g/dL (which can be maintained by blood transfusion).

   II.Liver function: the upper limit of the normal value of total bilirubin less than 1.5 times, the upper limit of normal value of alanine aminotransferase and glutamic pyruvic aminotransferase, less than 2.5 times the normal value, such as the liver metastasis and the upper limit of the normal value of the aminotransferase less than 5 times; Child-Pugh grade of liver function: A and a better B grade (less than 7); Barcelona Clinic Liver Cancer(BCLC)staging: B-C stage.

   III.Renal function: creatinine is less than 1.25 times the normal upper limit, and the creatinine clearance rate is more than 60ml/min.
9. Patients who adherence to research and follow-up procedures.
10. Patients who can understand and voluntarily sign informed consent.

Exclusion Criteria:

1. Patients with other malignant tumors over the last 5 years.
2. Patients who received chemotherapy, biotherapy or other anticancer drugs is less than 4 weeks.
3. Patients with the following and above conditions:

   I.Patients with symptomatic central nervous system metastases or spinal cord compression.

   II.Patients with peripheral neuropathy symptoms, grade NCI(National Cancer Institute)>gradeII.

   III.Patients with any unstable systemic disease (including active infection, poor control of hypertension,unstable angina,congestive heart failure, liver, kidney or metabolic diseases).

   IV.Patients with severe pulmonary interstitial changes, pulmonary fibrosis, and irreversible respiratory insufficiency.

   V.Patients who are not receiving oral administration, need high energy intravenous nutrition, have undergone previous operations affecting absorption, active gastrointestinal ulcer and chronic diarrhea.

   VI. Patients with serious, uncontrolled medical and infectious diseases. VII. Patients with severe electrolyte imbalance. VIII. Patients with diffuse intravascular coagulation. IX. Patients who known allergies to platinum and Everolimus targeted drugs
4. Patients with cognitive and psychological abnormality
5. Patients who use other test drugs or participate in other clinical trials.
6. Researchers believe that subjects may not be able to complete the study or may not be able to comply with the requirements of this study (for management or other reasons).

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 36 months
  Progression free survival of All the Evaluable Participants.Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0).(Note: the appearance of one or more new lesions is also considered progression).
OS | 36months
  Overall Survival of the Participants

SECONDARY OUTCOMES:
ORR | 36 months
  Objective Response Rate is defined as the proportion of patients with complete response(CR) or partial response(PR).
DCR | 36 months
  Disease control is defined as the proportion of patients who had a best response rating of complete response, partial response, or stable disease, and lasted at least 4 weeks.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Tianjin First Center Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No